CLINICAL TRIAL: NCT03945656
Title: A Trial Investigating the Hypoglycaemic Response to Overdosing of NNC0148-0287 C (Insulin 287) in Subjects With Type 2 Diabetes
Brief Title: A Research Study of How Overdosing of a New Once Weekly Medicine NNC0148-0287 C (Insulin 287) Influences the Blood Sugar Level in People With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4462; U1111-1214-2688 (Other: World Health Organization (WHO)); 2018-001993-74 (EudraCT Number)
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin 287 followed by insulin glargine (Experimental): Run-in period (3 to 28 days): Once daily insulin glargine treatment with or without any usual metformin treatment.
  After run-in, participants will receive insulin 287 once a week (OW) for 6 weeks.
  After insulin 287 treatment, participants will receive insulin glargine U100 OD for 12 days.
  Interventions: Drug: insulin icodec; Drug: Insulin glargine
- Insulin glargine followed by insulin 287 (Active Comparator): Run-in period (3 to 28 days): Once daily insulin glargine treatment with or without any usual metformin treatment.
  After run-in, participants will receive insulin glargine U100 OD for 12 days.
  After insulin glargine treatment, participants will receive insulin 287 OW for 6 weeks.
  Interventions: Drug: insulin icodec; Drug: Insulin glargine

INTERVENTIONS:
Drug: insulin icodec — Participants will receive subcutaneous (s.c.) injections of insulin 287 OW for 6 weeks
  Other Names: Insulin 287
Drug: Insulin glargine — Participants will receive daily s.c. injections of insulin glargine U100 for 12 days

SUMMARY:
This study is comparing the effect of a long-acting insulin analogue (insulin 287) with insulin glargine (Lantus®) in subjects with type 2 diabetes. In addition, the study is looking at symptoms of low blood sugar, awareness of low blood sugar and the time and amount of glucose needed to recover from low blood sugar after injecting 2 and 3 times the basal dose of insulin 287 and glargine. The purpose of the study is to make a once-weekly injectable basal insulin treatment for people with type 2 diabetes. Participants will get insulin 287 as well as insulin glargine - which treatment any participant gets first is decided by chance. Insulin 287 is a new medicine; insulin glargine can already be prescribed. The study medicines will be in a pen, and must be injected with a needle in the thigh once per day (insulin glargine) or once per week (insulin 287). The study will last for minimum 3 months and up to approximately 6 months. Participants will have 21 clinic visits and at least 2 phone calls with the study doctor. The participants' health will be monitored carefully and blood samples will be taken at the clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 18 and 72 years (both inclusive) at the time of signing informed consent.
* Body mass index between 18.5 and 37.9 kg/m^2 (both inclusive).
* Diagnosed with type 2 diabetes mellitus greater than or equal to 180 days prior to the day of screening.
* Glycosylated haemoglobin type A1c (HbA1c) less than or equal to 9.0% (less than or equal to 74 mmol/mol) at screening.
* Current total daily insulin treatment between 0.2 and 1.0 U/kg/day (both inclusive).

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological conditions (except conditions associated with diabetes mellitus).

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Clinically significant hypoglycaemia (Double dose): Clinically significant hypoglycaemia (Plasma glucose [PG] less than 3.0 mmol/L [54 mg/dL]) after 2 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 times the individualised optimal basal dose of insulin (day 17 for insulin 287, day 4 for insulin glargine) until termination of the clamp the following day
  Yes/No
  Blood sugar lower than 3.0 mmol/L (54 mg/dL) after receiving a double dose of basal insulin
  Number of subjects experiencing an event is to be reported

SECONDARY OUTCOMES:
PG (nadir) - PG concentration at nadir after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Measured in mmol/L
  Minimum blood sugar level achieved after receiving a double or triple dose of basal insulin
t (decline, PG 5.5 mmol/L - PG 3.0 mmol/L) - Time from start of hypoglycaemia induction until a PG concentration of 3.0 mmol/L (54 mg/dL) is reached after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Measured in hours
  Time from when blood sugar is normal [5.5 mmol/L (100 mg/dL)] until blood sugar is 3.0 mmol/L (54 mg/dL) after receiving a double or triple dose of basal insulin
t (decline, PG 5.5 mmol/L - PG nadir) - Time from start of hypoglycaemia induction until PGnadir is reached after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Measured in hours
  Time from when blood sugar is normal [5.5 mmol/L (100 mg/dL)] until blood sugar is at a minimum level after receiving a double or triple dose of basal insulin
t (recovery, PG nadir - PG 5.5 mmol/L) - Time to increase from PGnadir to a PG concentration of 5.5 mmol/L (100 mg/dL) after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Measured in hours
  Time from when blood sugar is at a minimum level until blood sugar is normal [5.5 mmol/L (100 mg/dL)] during recovery from low blood sugar after receiving a double or triple dose of basal insulin
C (glucagon, PG nadir) - Plasma glucagon concentration at PGnadir after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Measured in pg/mL
  Blood level of the glucagon hormone at the time point when blood sugar is at a minimum level after receiving a double or triple dose of basal insulin
C (adrenaline, PG nadir) - Plasma adrenaline concentration at PGnadir after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Measured in pg/mL
  Blood level of the adrenaline hormone at the time point when blood sugar is at a minimum level after receiving a double or triple dose of basal insulin
C (noradrenaline, PG nadir) - Plasma noradrenaline concentration at PGnadir after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Measured in pg/mL
  Blood level of the noradrenaline hormone at the time point when blood sugar is at a minimum level after receiving a double or triple dose of basal insulin
C (growth hormone [GH], PG nadir) - Serum growth hormone concentration at PGnadir after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Measured in ng/mL
  Blood level of GH at the time point when blood sugar is at a minimum level after receiving a double or triple dose of basal insulin
C (cortisol, PG nadir) - Serum cortisol concentration at PGnadir after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Measured in ng/mL
  Blood level of the cortisol hormone at the time point when blood sugar is at a minimum level after receiving a double or triple dose of basal insulin
Pulse (PG 5.5 mmol/L - PG nadir) - Change in pulse rate from a PG concentration of 5.5 mmol/L (100 mg/dL) until PGnadir after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Measured in beats/min
  Change in pulse from the time point when blood sugar is normal [5.5 mmol/L (100 mg/dL)] until the time point when blood sugar is at a minimum level after receiving a double or triple dose of basal insulin
Diastolic blood pressure (DBP) (PG 5.5 mmol/L - PG nadir) - Change in diastolic blood pressure from a PG concentration of 5.5 mmol/L (100 mg/dL) until PGnadir after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Measured in mmHg
  Change in DBP from the time point when blood sugar is normal [5.5 mmol/L (100 mg/dL)] until the time point when blood sugar is at a minimum level after receiving a double or triple dose of basal insulin
Systolic blood pressure (SBP) (PG 5.5 mmol/L - PG nadir) - Change in systolic blood pressure from a PG concentration of 5.5 mmol/L (100 mg/dL) until PGnadir after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Measured in mmHg
  Change in SBP from the time point when blood sugar is normal [5.5 mmol/L (100 mg/dL)] until the time point when blood sugar is at a minimum level after receiving a double or triple dose of basal insulin
Digit Symbol Substitution Test (DSST) (PG 5.5 mmol/L - PG nadir) - Change in DSST score from a PG concentration of 5.5 mmol/L (100 mg/dL) until PGnadir after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Number of correct responses
  Change in performance in the DSST (a cognitive ability test) from the time point when blood sugar is normal [5.5 mmol/L (100 mg/dL)] until the time point when blood sugar is at a minimum level after receiving a double or triple dose of basal insulin
Four-Choice Reaction Time (4CRT) (reaction 4CRT) (PG 5.5 mmol/L - PG nadir) - Change in 4CRT performance from a PG concentration of 5.5 mmol/L (100 mg/dL) until PGnadir after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Measured in msec
  Change in reaction time in the 4CRT test (a cognitive ability test) from the time point when blood sugar is normal [5.5 mmol/L (100 mg/dL)] until the time point when blood sugar is at a minimum level after receiving a double or triple dose of basal insulin
4CRT (% correct answers) (PG 5.5 mmol/L - PG nadir) - Change in 4CRT performance (% correct answers) from a PG concentration of 5.5 mmol/L (100 mg/dL) until PGnadir after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Measured in %-points
  Change in the percentage correct answers in the 4CRT test (a cognitive ability test) from the time point when blood sugar is normal [5.5 mmol/L (100 mg/dL)] until the time point when blood sugar is at a minimum level after receiving a double or triple dose of basal insulin
Trail Making B test (TMB) (PG 5.5 mmol/L - PG nadir) - Change in TMB from a PG concentration of 5.5 mmol/L (100 mg/dL) until PGnadir after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Measured in sec
  Change in performance in the TMB (a cognitive ability test) from the time point when blood sugar is normal [5.5 mmol/L (100 mg/dL)] until the time point when blood sugar is at a minimum level after receiving a double or triple dose of basal insulin
Hypoglycaemic symptoms score (HSS) (PG 5.5 mmol/L - PG nadir) - Change in HSS from a PG concentration of 5.5 mmol/L (100 mg/dL) to PGnadir after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Test score (arbitrary units)
  Change in symptoms of low blood sugar from the time point when blood sugar is normal [5.5 mmol/L (100 mg/dL)] until the time point when blood sugar is at a minimum level after receiving a double or triple dose of basal insulin
Hypoglycaemia awareness (HA) (PG nadir) - HA at PGnadir after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Yes/No
  Number of subjects with a feeling of low blood sugar at the time point when blood sugar is at a minimum level after receiving a double or triple dose of basal insulin
AUC (GIR, recovery, PG nadir -PG 5.5 mmol/L) - Area under the glucose infusion rate-time profile during recovery from PGnadir to a PG concentration of 5.5 mmol/L (100 mg/dL) after 2 and 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Measured in mg/kg
  Amount of glucose needed to be infused to increase blood sugar from a minimum level to a normal level [5.5 mmol/L (100 mg/dL)] during recovery from low blood sugar after receiving a double or triple dose of basal insulin
AUC (GIR, recovery, PG 5.5 mmol/L, 0-6h)-Area under the glucose infusion rate-time profile during 6 hours at a PG concentration of 5.5 mmol/L (100 mg/dL) after recovery from hypoglycaemia after 2 & 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 2 and 3 times the individualised optimal basal dose of insulin (day 17/day 38 for insulin 287, day 4/day 11 for insulin glargine) until termination of the clamp the following day
  Measured in mg/kg
  Amount of glucose needed to be infused to keep blood sugar at a normal level [5.5 mmol/L (100 mg/dL)] for 6 hours after recovery from low blood sugar after receiving a double or triple dose of basal insulin
Clinically significant hypoglycaemia (Triple dose) - Clinically significant hypoglycaemia [PG less than 3.0 mmol/L (54 mg/dL)], after 3 times the individualised optimal basal dose of insulin | From start of hypoglycaemia induction after 3 times the individualised optimal basal dose of insulin (day 38 for insulin 287, day 11 for insulin glargine) until termination of the clamp the following day
  Yes/No
  Blood sugar lower than 3.0 mmol/L (54 mg/dL) after receiving a triple dose of basal insulin
  Number of subjects experiencing an event is to be reported

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Background] Pieber TR, Arfelt KN, Cailleteau R, Hart M, Kar S, Mursic I, Svehlikova E, Urschitz M, Haahr H. Hypoglycaemia frequency and physiological response after double or triple doses of once-weekly insulin icodec vs once-daily insulin glargine U100 in type 2 diabetes: a randomised crossover trial. Diabetologia. 2023 Aug;66(8):1413-1430. doi: 10.1007/s00125-023-05921-8. Epub 2023 Jun 13. PMID 37308751